CLINICAL TRIAL: NCT06001879
Title: Protocol Title : Development, Validation, and Evaluation of the Effectiveness of Simulation in Basic Life Support Training (SBLST) on Newly Employed Nurses in Governmental Jordanian Hospitals.
Brief Title: The Study Focuses on Training Newly Employed Nurses With Two Groups Interventional (Simulation Training) & Control (Brochure) Group Using BLS -AHA 2020 Using Simulation, the Test Includes Pre-test & 2 Post-test Surveys to Assess Knowledge, Practice & Confidence Level.
Acronym: BLS-NEN-HCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: yousef Shukry Mohammad Abu-Wardeh (Other)
Responsible Party: Sponsor-Investigator, yousef Shukry Mohammad Abu-Wardeh, PHD STUDENTS aCUTE AND CRITICAL CARE IN NURSING, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JEPeM Code :USM/JEPeM/22110681
Record Dates: First submitted 2023-07-22; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy Nurses; Educational Activities
Keywords: pretest-post test and intervention

STUDY DESIGN:
Intervention Model Description: The study design is a basic experimental study design, randomized control trial (RCT) design, SBLST for the intervention group and standard intervention to the control group by using a brochure; the SBLST intervention among the control group was delayed until the end of data collection as an appreciation for their participation in the study, control group participants are wait-listed and exposed to the experimental treatment at a later point.
  Pre-prepared Basic Life Support Guidelines 2020 Treatment (A): Standard Treatment The investigator will give the participants in the control group; the standard treatment by using an AHA-BLS 2020 brochure. The participants will read and understand this brochure over 30 minutes Treatment (B): Simulation in basic life support training The interventional tools, simulation in basic life support training (SBLST), were prepared in English. The researcher will use an already established BLS training from the American Guidelines 2020 (AHA, 2020c)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBLST Group (Experimental): Treatment (B): Simulation in basic life support training The interventional tools, simulation in basic life support training (SBLST), were prepared in English. The researcher will use an already established BLS training from the American Guidelines 2020, a simplified two-part; PowerPoint presentation and clinical simulation training.
  Interventions: Other: Simulation in basic life support training (SBLST)
- Standard Group (Active Comparator): The investigator will give the participants in the control group; the standard treatment by using an AHA-BLS 2020 brochure. The participants will read and understand this brochure over 30 minutes, including a brief guideline about basic life support guidelines, and after these 30 minutes, the participants will move to the post-test.
  Interventions: Other: standard treatment by using an AHA-BLS 2020 brochure

INTERVENTIONS:
Other: Simulation in basic life support training (SBLST) — The interventional tools, simulation in basic life support training (SBLST), were prepared in English. The researcher will use an already established BLS training from the American Guidelines 2020, a simplified two-part; PowerPoint presentation, and clinical simulation training.
  Arms: SBLST Group
Other: standard treatment by using an AHA-BLS 2020 brochure — The participants will read and understand this brochure over 30 minutes, including a brief guideline about basic life support guidelines, and after these 30 minutes, the participants will move to the post-test
  Arms: Standard Group

SUMMARY:
The general objective of this study is to develop, validate and evaluate the effectiveness of simulation in basic life support training (SBLST) among newly employed nurses in Jordanian governmental hospitals; the study design is a basic experimental study design, randomized control trial (RCT) design, the dependant variables measure in this study; knowledge, practice and confidence by using a pre-test and two follow up tests, two groups are participating in this study; experimental and control group. The control group treatment is the standard intervention (brochure), and the experimental group intervention is a simulation in basic life support training (SBLST). The study process includes four steps

* Perform the pre-test (assess knowledge, practice confidence surveys
* Education intervention knowledge and practice
* Perform the post-test 1 (assess knowledge, practice confidence surveys
* Perform post-test 2 (assess knowledge, practice confidence surveys

DETAILED DESCRIPTION:
The general objective of this study is to develop, validate and evaluate the effectiveness of simulation in basic life support training (SBLST) among newly employed nurses in Jordanian governmental hospitals; the study design is a basic experimental study design, randomized control trial (RCT) design, the dependant variables measure in this study; knowledge, practice and confidence by using a pre-test and two follow up tests, two groups are participating in this study; experimental and control group. The control group treatment is the standard intervention (brochure), and the experimental group intervention is a simulation in basic life support training (SBLST); researchers' hypothesized that there are no significant differences between the control and experimental group in the inclusion criteria and pre-test score; furthermore, the simulation in basic life support training intervention significantly improves knowledge, practice and confidence level among newly employed nurses (NEN) in Jordanian governmental hospitals; moreover, the is a significant difference between control and experimental group in the post-test scores in all dependant variables. The study process include four steps

* Perform the pre-test (assess knowledge, practice confidence surveys
* Education intervention knowledge and practice
* Perform the post-test 1 (assess knowledge, practice confidence surveys
* Perform post-test 2 (assess knowledge, practice confidence surveys

Study title:

DEVELOPMENT, VALIDATION, AND EVALUATION OF THE EFFECTIVENESS OF SIMULATION IN BASIC LIFE SUPPORT TRAINING (SBLST) ON NEWLY EMPLOYED NURSES IN GOVERNMENTAL JORDANIAN HOSPITALS

Research Hypotheses i. The simulation in basic life support training intervention effectively improves knowledge among newly employed nurses (NEN) in Jordanian governmental hospitals.

ii. The simulation in basic life support training intervention effectively improves practice among newly employed nurses (NEN) in Jordanian governmental hospitals.

iii. The simulation in basic life support training intervention effectively improves the confidence level among newly employed nurses (NEN) in Jordanian governmental hospitals.

iv. There is no significant difference in means between the pre-test among the newly employed nurses (NEN) among interventional and the control groups in all dependent variables.

v. There is a significant mean difference between PRE-SBLST and all POST-SBLST results among NEN in all dependent variables.

Study Design The study design was a prospective, longitudinal, single-blind basic experimental design, randomized control trial (RCT) design.

Study Location The study was carried out in Jordan, Amman and Al-Zarqa City. The accessible population was NEN in five hospitals. The researchers selected three Jordanian hospitals. The selection was according to the capacity, capability of the institution and eligibility criteria. Computer-generated randomization (Random Allocation Software, version 1.0) was applied in blocks to allocate the hospitals by distributing them into two arms. The first arm was the control group; selected from three hospitals; Prince Hamza Hospital, AL-Basheer Hospital, and AL-Zarqa Governmental Hospital (n=51); the second arm was the interventional group from two hospitals; Prince Faisal Governmental Hospital and Dr.Jameel AL-Totanji Hospital.

Randomization of the Hospitals To prevent data contamination between the control and interventional groups, computer-generated randomization (Random Allocation Software, version 1.0) was applied in blocks to allocate the hospitals by distributing them into two arms. The first arm was the control group; selected from three hospitals; Prince Hamza Hospital, AL-Basheer Hospital, and AL-Zarqa Governmental Hospital (n=51); the second arm was the interventional group from two hospitals; Prince Faisal governmental hospital and Dr.Jameel AL-Totanji hospital. The control and interventional groups were selected from different hospitals because the researchers are always worried about data contamination and try to minimize it between the control and intervention groups; if the sample was selected from the same area and both groups worked closely together, the data would be contaminated.

The study consists of a pre-test, intervention, immediate post-test-1 after the intervention, and post-test-2 three months after the intervention. This study measured knowledge, practice, and confidence through pre- and post-tests in control and experimental groups. This study used two interventions: SBLST for the interventional group and AHA-BLS 2020 brochure as a standard treatment for the control group. Data collection proceeded using the Google Form Platform (A web-based instrument Copyrighted by Google application).

The evaluation process includes a pre-test and two follow-up assessments to measure knowledge, practice and confidence. The researcher will analyze the means of each test; the total dependent variables were 30 questions.

Research Instruments

Languages of the Tools According to the HCP educational level, all four sections of the tools assessment are written in English; furthermore, the researchers' assistance clarified any misunderstanding points or need for translation to the participants.

Tools Sections The tools consist of five sections; research information sheet and consent forms, demographical data, knowledge assessment tools, skills assessment tools, and confidence level assessment tools.

Research information sheet and Consent Forms The research information sheet is a piece of brief researcher information and contact details; it also includes subject information and a consent form with an area for the participant's signature when they are approved to participate in this study. Furthermore, the research information sheets include a participant's publication consent form.

Demographical data Demographic parts are attached; these data consist of dichotomous questions (Yes\NO), nominal data, ordinal data, and interval measurement questions. Nominal measurements include sex and ordinal assessment as educational level and area of experience; interval assessment questions include age and work experience. Dichotomous assessments (Yes\NO), asking if the participant previously participated in a CPR episode or observed any CPR before, if the participants had finished training the BLS using simulation previously, and if the participant gained the certification of BLS training from formal and accredited institutions.

Knowledge and practice Nursing knowledge is the interaction of science and research to improve practice. Researchers use a 13-question MCQ tool to assess knowledge. Nursing practice is performing the knowledge learned before; the researchers assessed skills using a tool consisting of ten MCQ. The participants got zero for each wrong answer and one mark for each correct answer.

Confidence Confidence is the building and accomplishment of the nursing profession through knowledge acquisition, skills, and critical thinking. Confidence is the positive feeling of faith and dependability to perform BLS without fear and free from risk to the patient. The researchers assessed confidence level using seven statements rated as a dropdown in percent value from the lowest value of 5% to the highest value of 100%.

Study process steps

1. Pre-test After NEN enrolled according to the inclusion criteria for both the control group and experimental group (n= 102), the participants started by signing the informed consent, filled out the demographical data and pre-test as proactive steps before the intervention; many sessions of pre-test data collection and intervention were performed according to the availability of NEN, the arrangement of the hospital's nursing director. The estimated time to fill in the demographical data and pre-test is around 30 minutes. Oermann et al. (2020) addressed that the trainer performs a pre-test assessment to assess the effectiveness of SBLST. The investigators discussed the purpose of the study with the control group and explained to them the procedure to prevent any data contamination and minimize the interpretation of the survey content by the other research assistants.
2. Intervention The control group read the brochure containing a brief guideline about basic life support for 30-60 minutes before taking the post-test. Standard treatment ran from Dec 2022 to Jan 2023. One full day for SBLST intervention, from 5 to 7 hours for SBLST intervention, is required based on the recent research and uses AHA-2020 guidelines. The number of participants was ten NEN in each session. The interventional treatment consists of theoretical and practical parts. The SBLST intervention was conducted in an educational lab according to the hospital's capability; SBLST ran for seven days, from 22 Nov 2022 to 20-Dec, 2022.

   Researchers combined two frameworks in the SBLST. Miller's Pyramid and Kolb's Cycle; Miller's Pyramid focuses on teaching theoretical and practical aspects of the task through simulation and allowing trainees to perform the procedure independently with guidance; Kolb's Cycle suggests giving learners a scenario to practice until they eliminate errors before moving to another scenario. The SBLST intervention was reviewed by three experts in BLS and approved by the Jordanian Ministry of Health-Life Support Center. It was found to be compliant, safe and covered all aspects of AHA-2020. English experts provided feedback to improve clarity. A pilot study was conducted on 20 nurses to calculate SBLST time, identify errors, monitor the progress and calculate Cronbach's Alpha.A pilot study was performed to check the stability of the tools. Cronbach's alpha of knowledge and skills assessment tools was 0.748, reflecting the suitability and strength of using these tools. Moreover, Cronbach's alpha of confidence tools was 0.731, reflecting the suitability and stability of the confidence tools.

   Adult half-body manikin and a pediatric full-body manikin are necessary; with lung bag inflation and deflation characteristics, palpable carotid pulse, the chest includes spring inside to facilitate chest recoil, and chest compression board, bag-valve-mask-ventilation, chest compression performed on the Charlie simulator to relieve choking. The principles investigator (PI) had a master's degree in critical care nursing, eighteen years of experience between ICUs, lecturers and clinical instructors, valid BLS and ACLS, training of trainers in nursing education, and randomized control trial training. The facilitator must have CPR certifications in BLS and ACLS, enough expertise in education and training, and good communication skills. The investigator had a master's degree in critical care. Two research assistants supported the PI in collecting data; one research assistant for the control group and the other for the interventional group.
3. post-test All participants completed the immediate post-test-1 after the interventions. The post-tets-2 was conducted by providing the participants with a Google Form Platform link through their phone and email addresses. The post-test after three months evaluates whether the participants' level stayed at the same level or minimized by comparing the mean value between all post-tests. Forty-eight participants in the experimental group completed post-test-2 with a response rate of 94%, and 45 participants in the control group with a response rate of 88%.

Sample Size Estimation Sample size calculation is performed by using G*POWER software (version 3.1); sample size calculation is summarized and consists of the following steps (1) Select the test family (F-test family), (2) Select the statistical test (Select ANOVA-repeated test, between factors), the preliminary test analysis the researchers used in this study, the rationale for using the Select ANOVA-repeated test between factors due to measuring many dependent variables means at different time points. (3) The parameters selected to calculate sample size include one side tail, alpha (α) and equals (0.05)- type one error, Power (P) and equal (0.8), effect size, the number of groups is two (each group = n\2) n= the estimated sample size, number of measurements were four measurements (Pre-test, Post-test immediately, Post-test after two months, and Post-test after three months).

Effect Size (ES) = 0.26, automatically calculated by G*Power software, depending on the sample size of the previous study, the effect size is calculated, the Control group's post-test result M±SD was equal (25.03±3.04) with a sample size of 28 participants, and the interventional group (26.64±2.64) with sample size 29 participants. The sample size is 72 participants; because the research study continued for three months, the invistigators added a 10% drop rate for each month, so the drop rate is 30%. Final sample size estimation including drop rate (n\1-dropout rate) = 72/(1-0.30) = 102 participants, the intervention group arm is 51 participants, and The largest sample size was obtained from the interventional group, more than the Control Group and the Control group arm 51 participants.

Simple Random Sampling of the Participants After obtaining ethical approval and permission to conduct the study from the Ministry of Health in Jordan, approval letter (Education/Info\ 15177) and ethical approval letter (MOH/REC/2022/340), The researchers started the formal face-to-face visits to arrange with the nursing director and a continuous education office in the selected hospitals about the study objective and how the study would proceed; The researchers received the activation letter to initiate the study and prepared the list of the available participants who met the study's eligibility criteria. The number of participants depends on the availability of newly employed nurses in the institution who meet the inclusion criteria. The researchers randomly selected the participants from the participants' list by randomly sampling from newly employed nurses in each hospital for interventional and control groups.

. The response of the control group hospitals was as the following; the nursing director and continuous education in AL-Zarqa Governmental Hospital responded by providing all the information about participants and selecting a time and day to perform the Pre-test, standard treatment and the immediate post-test. Prince Hamzah Hospital and AL-Basheer Hospital gave the researcher the names of departments in the hospital, including those with NEN, and the invistigators visited these departments to select the available NEN randomly and performed Pre-test, standard treatment, and immediate post-test in their departments.

The response of the interventional group hospitals was as the following; Prince Faisal Governmental Hospital and Dr.Jameel AL-Totanji Hospital scheduled many days and times to perform the intervention, and the hospitals arranged with the available participants who met the eligibility criteria; then, the researcher selected the participants randomly.

Ethical Considerations

1. Permission to Conduct the Study Regarding ethical considerations, approval for the study was obtained from the Human Research Ethics Committee (HREC), Universiti Sains Malaysia (USM). Moreover, ethical approvals to initiate SBLST intervention in Jordanian Hospitals in Amman and AL-Zarqa city were obtained from the Ministry of Health in Jordan; the study protocol was revised and approved for implementation by Jawatankuasa Etika Penyilidikan Manusia Universiti Sains Malaysia (JEPeM-USM) with study protocol code USM/JEPeM/22110681, which compliance with the Declaration of Helsinki, International Conference on Harmonization (ICH) Guidelines, Good Clinical Practice (GCP) Standards, Council for International Organizations of Medical Sciences (CIOMS) Guidelines, World Health Organization (WHO) Standards and Operational Guidance for Ethics Review of Health-Related Research and Surveying and Evaluating Ethical Review Practices, EC/IRB Standard Operating Procedures (SOPs), and Local Regulations and Standards in Ethical Review.
2. Subject Vulnerability There is no vulnerability group in this study. All the participants were nurses over 20 years old and working in hospitals; no participants had handicaps or physical problems. The participants made the voluntary choice to take part in the trial. The researchers discussed the study's objectives, methods, benefits and risks. The study was free from any potential hazards or adverse effects on participants, no intervention was applied in emergencies, and no medicine product will be used in this study. The procedure was simple, the devices used in the intervention were safe, and the investigator was instructed to frequently ask the participant about health and physical condition, especially during chest compression.

   The participants who signed a hard copy of the consent are part of this trial study. During all study phases, the participants will be asked using the electronic method; Google Form Platform, if they would like to participate in this study, and they will answer (YES\NO) before completing the questionnaires. Furthermore, the intervention will be applied in simulation; the participant voluntarily withdraws from the study without any influence or effect on annual evaluation or salary. The institutions took full responsibility for the trial and protecting the participants and treated the participants if there were unexpected adverse effects or physical harm.

   The research includes minimal risk toward participants, observable by the time length and components of the intervention; participants may be feeling discomfort. This risk is equal to the nurses' daily life activity. They can be adapted with this minimal risk; only four components require a long time to cover the knowledge and practice in the intervention, but the other four components are easy and need a short time. The researchers planned to minimize the participant's discomfort due to the time and length of the intervention by giving the participant "break times" between the components of the intervention.
3. Declaration of Absence of Conflict of Interest The researchers had declared that there was no conflict of interest, and all co-authors had no financial interest to report. The invistigators certify that the first author is purely a Ph.D. student's original work and has not been given to submit to other universities or journals.
4. Privacy and Confidentiality When the study was completed, the trial master files and documents were protected and kept safe, and all records were kept confidential. Furthermore, the data collected is not associated with individuals by name but only by phone number and email to contact them later to complete the post-test; data is kept properly and handled only in the research. In addition, the researchers also emphasized that only research groups can access the relevant data in this research and not use it in the future without consent from the participants; moreover, after finishing the study, the data will archive properly according to the policy.
5. Community Sensitivities and Benefits The intervention benefits of NEN as a part of a contentious education, and the knowledge and practice shared through the natural learning process in the classroom, face-to-face learning, and the questionnaires filled using an electronic method, Google Forms Platform; there is no sensitive information about the participants. The primary benefits of this study's findings toward participants are to increase newly employed nurses' knowledge, practice skills, and confidence level when facing critical situations inside or outside the hospitals, increases professionalism in all healthcare delivery systems, self-esteem, improve newly employed nurses' performance competency, decision-making, satisfaction, to decrease turnovers and dissatisfaction. Furthermore, the benefits of this study are to develop patient care processes and enhance the victims' survival and patient satisfaction, maintain patient safety, enhance the welfare and hospital discharge outcomes, become cost-effective for patients and their families, and keep patients away from hazards.
6. Incentive and Reimbursement The researcher verbally thanked all participants for their sincere cooperation following the completion. Furthermore, the researcher planned to give the control group an SBLST on a selected day; finally, the participant received feedback about the pre and post-result and a certification attendance of 4 hours from the researcher, adding to the required job development hours in the yearly self-evaluation form.
7. Collaborative Study Terms of Reference: None

ELIGIBILITY:
Inclusion Criteria The researchers tried to maintain homogeneity and minimize any variations among the participants by

1. selecting both interventional and control groups from newly employed nurses
2. Male and female participants
3. Participants only who understand the questionnaires and interventions in English
4. Participants who were previously on-seat undergraduate nursing students last two years, 2020 (4th year nursing bachelor level) and 2021 (3rd year nursing bachelor level) in the period of the COVID-19 pandemic and received basic and clinical learning by online method, and now became a newly employed nurse (NEN) in hospitals and delivered care to the patient.
5. Participants can attend five to seven hours of SBLST sessions.
6. For more control, we selected nurses who rarely face CPR and do not attend BLS raining the last two years.

Exclusion Criteria

1. The researchers excluded the NEN participants working in intensive care units because ICU nurses face CPR and perform BLS daily.
2. Excluded participants with medical or physical health problems (e.g., pregnant women and participants complaining of lower back pain).
3. Participants who attended CPR training less than two years previously were also excluded. Finally,
4. NEN who upgraded their educational degree from a diploma to a bachelor's degree were excluded.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The Effectiveness of Simulation in basic life support training (SBLST) on the Knowledge Score | 6 Months after finish all data collection
  To evaluate the effectiveness of SMBST on knowledge scores, investigators will conduct three measurements: a pretest, an immediate post-test after the intervention, and a post-test 2 after three months for both experimental and control groups. Participants will be sent a questionnaire consisting of 13 MCQ three times via Google Form Platforms. These questions will be sent to their cell phone numbers. Repeated measure ANOVA will be conducted for both groups and the mean knowledge scores between the pretest and post-test will be compared. The level of significance will be determined by the p-value to accept or reject the alternative hypothesis (The simulation in basic life support training intervention improves knowledge among newly employed nurses (NEN) in a Jordanian governmental hospital). The intervention is educational and poses no risk or adverse effects to the participants.
The Effectiveness of Simulation in basic life support training (SBLST) on the Practice Score | 6 moths after finish all data collection
  The investigators performed three measurements to assess the effectiveness of SMBST on practice score; Pretest, immediate-posttest after the intervention, and post-test-2 after three months of the intervention for both experimental and control groups. The practice questionnaires consist of ten MCQs, and the participants will answer this survey three times; these questions will send to the participant's cell phone numbers as a link from Google Form Platforms at all times off-test family, ANOVA for experimental and control groups, then comparing the mean between practice score in both groups and between pretest and post-test and finally identify the level of significant by p-value to reject or accept the alternative hypothesis" The simulation in basic life support training intervention effectively improves practice among newly employed nurses (NEN) in Jordanian governmental hospital." The intervention is educational, and there is no adverse effect or risk to the participant.
The Effectiveness of Simulation in basic life support training (SBLST) on the Confidence Level | 6 moths after finish all data collection
  The effectiveness of SMBST on confidence levels will be assessed by measuring pretest, immediate posttest, and post-test-2 results for both experimental and control groups. Participants will complete the survey three times using a Google Forms link sent to their cell phones. Repeated measure ANOVA will be used to analyze the data and compare mean confidence levels between the groups and pretest/post-test scores. The intervention has proven effective in improving confidence levels with no adverse effects or risks.

SECONDARY OUTCOMES:
There are no significant differences between the control and experimental groups in the knowledge score pretest | 2 month after finsh the pre-test of both group
  Before implementing any interventions for the experimental and control groups, the investigator ensures that the pretest levels of both groups are significantly similar to ensure accurate measurement. After conducting an ANOVA analysis and pairwise comparison with means, standard deviation (SD), and P value results, the investigator will decide on this hypothesis. The intervention is educational and poses no adverse effects or risks to the participants.
There are no significant differences between the control and experimental groups in the practice score pretest | 2 month after finsh the pre-test of both group
  Before implementing any interventions for the experimental or control groups, the investigator takes measures to ensure that both groups possess comparable pretest scores, thus guaranteeing precise measurements. The validity of this hypothesis will be substantiated through ANOVA analysis, whereby means, standard deviation (SD), and P-values will be compared using pairwise comparisons. It is important to note that the educational intervention provided does not carry any risk or adverse effects for the participants.
There are no significant differences between the control and experimental groups in the pretest regarding confidence level. | 2 month after finsh the pre-test of both group
  Before performing any intervention for the intervention; and experimental groups, the investigator makes sure that the pretest of both groups is significantly the same level to ensure the accuracy of the measurement; the investigator will decide on this hypothesis after ANOVA analysis and use pairwise comparison with means, standard deviation (SD), and P value results. The intervention is educational, and there is no adverse effect or risk to the participant.
Significant differences exist between the control and experimental groups in the post-tests on knowledge scores. | 6 moths after finish all data collection
  The investigator will assess the effectiveness of SBLST on the experimental group by comparing post-test mean and SD and assess the level of significance (p-value) for the control and experimental group to decide that the SBLST was effective on knowledge score using ANOVA repeated measure analysis. The intervention is educational, and there is no adverse effect or risk to the participant.
Significant differences exist between the control and experimental groups in the post-test after the interventions on practice score | 6 moths after finish all data collection
  The investigator will assess the effectiveness of SBLST on the experimental group by comparing post-test mean and SD and assess the level of significance (p-value) for the control and experimental group to decide that the SBLST was effective on practice score using ANOVA repeated measure analysis. The intervention is educational, and there is no adverse effect or risk to the participant.
Significant differences exist between the control and experimental groups in the post-test after the interventions on the confidence level | 6 moths after finish all data collection
  The investigator will assess the effectiveness of SBLST on the experimental group by comparing post-test mean and SD and assess the significance level (p-value) for the control and experimental group to decide that the SBLST was effective on confidence level using ANOVA repeated measure analysis. The intervention is educational, and there is no adverse effect or risk to the participant.

OTHER OUTCOMES:
There are no differences between the control and experimental groups in the inclusion criteria | 2 month after finsh the pre-test of both group
  The investigators selected inclusion criteria for both the control and experimental group, and both groups should be Homogenous in the demographical data by using Mann-Witney U-test and checking the median and IQ range. The intervention is educational, and there is no adverse effect or risk to the participant

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of Health, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Only the participant data related to the study after participate and publication consent without mentioned name, ID, email...and providing the privacy
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after finish and publish the study and will not use in any other study
Access Criteria: Data is kept properly and handled only in the research. In addition, the researchers also emphasized that only research groups can access the relevant data in this research and not use it in the future without consent from the participants; moreover, after finishing the study, the data will archive properly according to the policy.

REFERENCES:
- [Background] Pallas JD, Smiles JP, Zhang M. Cardiac Arrest Nurse Leadership (CANLEAD) trial: a simulation-based randomised controlled trial implementation of a new cardiac arrest role to facilitate cognitive offload for medical team leaders. Emerg Med J. 2021 Aug;38(8):572-578. doi: 10.1136/emermed-2019-209298. Epub 2021 Jan 26. PMID 33500268
- [Background] Nolan JP, Ornato JP, Parr MJA, Perkins GD, Soar J. Resuscitation highlights in 2019. Resuscitation. 2020 Mar 1;148:234-241. doi: 10.1016/j.resuscitation.2020.02.001. Epub 2020 Feb 7. No abstract available. PMID 32044335
- [Background] Zhou XL, Wang J, Jin XQ, Zhao Y, Liu RL, Jiang C. Quality retention of chest compression after repetitive practices with or without feedback devices: A randomized manikin study. Am J Emerg Med. 2020 Jan;38(1):73-78. doi: 10.1016/j.ajem.2019.04.025. Epub 2019 Apr 12. PMID 31005392
- [Result] Al Gharibi Msn KA, Arulappan MSc N PhD DNSc J. Repeated Simulation Experience on Self-Confidence, Critical Thinking, and Competence of Nurses and Nursing Students-An Integrative Review. SAGE Open Nurs. 2020 Jun 1;6:2377960820927377. doi: 10.1177/2377960820927377. eCollection 2020 Jan-Dec. PMID 33415282
- [Result] Abelsson A, Odestrand P, Nygardh A. To strengthen self-confidence as a step in improving prehospital youth laymen basic life support. BMC Emerg Med. 2020 Jan 30;20(1):8. doi: 10.1186/s12873-020-0304-8. PMID 32000691
- [Result] Aksoy ME. Comparing Basic Life Support Serious Gaming Scores With Hands-on Training Platform Performance Scores: Pilot Simulation Study for Basic Life Support Training. JMIR Serious Games. 2020 Nov 25;8(4):e24166. doi: 10.2196/24166. PMID 33237035
- [Result] Lott C, Truhlar A, Alfonzo A, Barelli A, Gonzalez-Salvado V, Hinkelbein J, Nolan JP, Paal P, Perkins GD, Thies KC, Yeung J, Zideman DA, Soar J; ERC Special Circumstances Writing Group Collaborators. European Resuscitation Council Guidelines 2021: Cardiac arrest in special circumstances. Resuscitation. 2021 Apr;161:152-219. doi: 10.1016/j.resuscitation.2021.02.011. Epub 2021 Mar 24. PMID 33773826
- [Result] Aliyari S, Pishgooie AH, Abdi A, Mazhari MS, Nazari MR. Comparing two teaching methods based on concept map and lecture on the level of learning in basic life support. Nurse Educ Pract. 2019 Jul;38:40-44. doi: 10.1016/j.nepr.2019.05.008. Epub 2019 May 31. PMID 31176242
- [Result] Armstrong P, Peckler B, Pilkinton-Ching J, McQuade D, Rogan A. Effect of simulation training on nurse leadership in a shared leadership model for cardiopulmonary resuscitation in the emergency department. Emerg Med Australas. 2021 Apr;33(2):255-261. doi: 10.1111/1742-6723.13605. Epub 2020 Aug 27. PMID 32856402
- [Result] Banfai B, Musch J, Betlehem J, Santa E, Horvath B, Nemeth D, Banfai-Csonka H. How effective are chest compressions when wearing mask? A randomised simulation study among first-year health care students during the COVID-19 pandemic. BMC Emerg Med. 2022 May 8;22(1):82. doi: 10.1186/s12873-022-00636-2. PMID 35527256
- [Result] Barakat M, Farha RA, Muflih S, Al-Tammemi AB, Othman B, Allozi Y, Fino L. The era of E-learning from the perspectives of Jordanian medical students: A cross-sectional study. Heliyon. 2022 Jul 11;8(7):e09928. doi: 10.1016/j.heliyon.2022.e09928. eCollection 2022 Jul. PMID 35874065
- [Result] Borggreve AS, Meijer JMR, Schreuder HWR, Ten Cate O. Simulation-based trauma education for medical students: A review of literature. Med Teach. 2017 Jun;39(6):631-638. doi: 10.1080/0142159X.2017.1303135. Epub 2017 Mar 30. PMID 28355934
- [Result] Binkhorst M, van der Aar IM, Linders M, van Heijst AFJ, de Boode WP, Draaisma JMT, Hogeveen M. Training practices in neonatal and paediatric life support: A survey among healthcare professionals working in paediatrics. Resusc Plus. 2021 Jan 6;5:100063. doi: 10.1016/j.resplu.2020.100063. eCollection 2021 Mar. PMID 34223335
- [Result] Bottiger BW, Lockey A, Aickin R, Bertaut T, Castren M, de Caen A, Censullo E, Escalante R, Gent L, Georgiou M, Kern KB, Khan AMS, Lim SH, Nadkarni V, Nation K, Neumar RW, Nolan JP, Rao SSCC, Stanton D, Toporas C, Wang TL, Wong G, Perkins GD. Over 675,000 lay people trained in cardiopulmonary resuscitation worldwide - The "World Restart a Heart (WRAH)" initiative 2018. Resuscitation. 2019 May;138:15-17. doi: 10.1016/j.resuscitation.2019.02.033. Epub 2019 Mar 2. No abstract available. PMID 30836172
- [Result] Bukiran A, Erdur B, Ozen M, Bozkurt AI. Retention of nurses' knowledge after basic life support and advanced cardiac life support training at immediate, 6-month, and 12-month post-training intervals: a longitudinal study of nurses in Turkey. J Emerg Nurs. 2014 Mar;40(2):146-52. doi: 10.1016/j.jen.2012.08.011. Epub 2013 Jan 7. No abstract available. PMID 23305947
- [Result] Semeraro F, Greif R, Bottiger BW, Burkart R, Cimpoesu D, Georgiou M, Yeung J, Lippert F, S Lockey A, Olasveengen TM, Ristagno G, Schlieber J, Schnaubelt S, Scapigliati A, G Monsieurs K. European Resuscitation Council Guidelines 2021: Systems saving lives. Resuscitation. 2021 Apr;161:80-97. doi: 10.1016/j.resuscitation.2021.02.008. Epub 2021 Mar 24. PMID 33773834
- [Result] Soar J, Bottiger BW, Carli P, Couper K, Deakin CD, Djarv T, Lott C, Olasveengen T, Paal P, Pellis T, Perkins GD, Sandroni C, Nolan JP. European Resuscitation Council Guidelines 2021: Adult advanced life support. Resuscitation. 2021 Apr;161:115-151. doi: 10.1016/j.resuscitation.2021.02.010. Epub 2021 Mar 24. PMID 33773825
- [Result] Charlier N, Van Der Stock L, Iserbyt P. Comparing student nurse knowledge and performance of basic life support algorithm actions: An observational post-retention test design study. Nurse Educ Pract. 2020 Feb;43:102714. doi: 10.1016/j.nepr.2020.102714. Epub 2020 Feb 19. PMID 32109754
- [Result] Christmals CD, Gross J, Aziato L, Armstrong SJ. The State of Nursing Research in Ghana: An Integrative Literature Review. SAGE Open Nurs. 2018 Nov 18;4:2377960818783820. doi: 10.1177/2377960818783820. eCollection 2018 Jan-Dec. PMID 33415196
- [Result] Costa IKF, Tiburcio MP, Costa IKF, Dantas RAN, Galvao RN, Torres GV. Development of a virtual simulation game on basic life support. Rev Esc Enferm USP. 2018 Nov 1;52:e03382. doi: 10.1590/S1980-220X2017047903382. English, Portuguese. PMID 30403269
- [Result] Couloures KG, Allen C. Use of Simulation to Improve Cardiopulmonary Resuscitation Performance and Code Team Communication for Pediatric Residents. MedEdPORTAL. 2017 Mar 16;13:10555. doi: 10.15766/mep_2374-8265.10555. PMID 30800757
- [Result] Curl ED, Smith S, Ann Chisholm L, McGee LA, Das K. Effectiveness of Integrated Simulation and Clinical Experiences Compared to Traditional Clinical Experiences for Nursing Students. Nurs Educ Perspect. 2016 Mar-Apr;37(2):72-7. PMID 27209864
- [Result] Requena-Mullor MDM, Alarcon-Rodriguez R, Ventura-Miranda MI, Garcia-Gonzalez J. Effects of a Clinical Simulation Course about Basic Life Support on Undergraduate Nursing Students' Learning. Int J Environ Res Public Health. 2021 Feb 3;18(4):1409. doi: 10.3390/ijerph18041409. PMID 33546328
- [Result] Dick-Smith F, Power T, Martinez-Maldonado R, Elliott D. Basic Life Support Training for undergraduate nursing students: An integrative review. Nurse Educ Pract. 2021 Jan;50:102957. doi: 10.1016/j.nepr.2020.102957. Epub 2020 Dec 22. PMID 33421680
- [Result] Ekert JO, Luchesa Smith A, Ramsey CL, Robinson N, Love J, Gothard P, Armitage AJ. Medical student-led simulation in COVID-19 crisis. Clin Teach. 2021 Jun;18(3):252-257. doi: 10.1111/tct.13308. Epub 2020 Dec 6. PMID 33280253
- [Result] Elgohary M, Palazzo FS, Breckwoldt J, Cheng A, Pellegrino J, Schnaubelt S, Greif R, Lockey A. Blended learning for accredited life support courses - A systematic review. Resusc Plus. 2022 May 10;10:100240. doi: 10.1016/j.resplu.2022.100240. eCollection 2022 Jun. PMID 35592876
- [Result] Garcia-Suarez M, Mendez-Martinez C, Martinez-Isasi S, Gomez-Salgado J, Fernandez-Garcia D. Basic Life Support Training Methods for Health Science Students: A Systematic Review. Int J Environ Res Public Health. 2019 Mar 3;16(5):768. doi: 10.3390/ijerph16050768. PMID 30832440
- [Result] Gonzalez-Salvado V, Rodriguez-Ruiz E, Abelairas-Gomez C, Ruano-Ravina A, Pena-Gil C, Gonzalez-Juanatey JR, Rodriguez-Nunez A. Training adult laypeople in basic life support. A systematic review. Rev Esp Cardiol (Engl Ed). 2020 Jan;73(1):53-68. doi: 10.1016/j.rec.2018.11.013. Epub 2019 Feb 23. English, Spanish. PMID 30808611
- [Result] Goodloe JM, Topjian A, Hsu A, Dunne R, Panchal AR, Levy M, McEvoy M, Vaillancourt C, Cabanas JG, Eisenberg MS, Rea TD, Kudenchuk PJ, Gienapp A, Flores GE, Fuchs S, Adelgais KM, Owusu-Ansah S, Terry M, Sawyer KN, Fromm P, Panczyk M, Kurz M, Lindbeck G, Tan DK, Edelson DP, Sayre MR. Interim Guidance for Emergency Medical Services Management of Out-of-Hospital Cardiac Arrest During the COVID-19 Pandemic. Circ Cardiovasc Qual Outcomes. 2021 Jul;14(7):e007666. doi: 10.1161/CIRCOUTCOMES.120.007666. Epub 2021 Jun 23. No abstract available. PMID 34157848
- [Result] Grasner JT, Herlitz J, Tjelmeland IBM, Wnent J, Masterson S, Lilja G, Bein B, Bottiger BW, Rosell-Ortiz F, Nolan JP, Bossaert L, Perkins GD. European Resuscitation Council Guidelines 2021: Epidemiology of cardiac arrest in Europe. Resuscitation. 2021 Apr;161:61-79. doi: 10.1016/j.resuscitation.2021.02.007. Epub 2021 Mar 24. PMID 33773833
- [Result] Greif R, Lockey A, Breckwoldt J, Carmona F, Conaghan P, Kuzovlev A, Pflanzl-Knizacek L, Sari F, Shammet S, Scapigliati A, Turner N, Yeung J, Monsieurs KG. European Resuscitation Council Guidelines 2021: Education for resuscitation. Resuscitation. 2021 Apr;161:388-407. doi: 10.1016/j.resuscitation.2021.02.016. Epub 2021 Mar 24. PMID 33773831
- [Result] Gutierrez-Puertas L, Garcia-Viola A, Marquez-Hernandez VV, Garrido-Molina JM, Granados-Gamez G, Aguilera-Manrique G. Guess it (SVUAL): An app designed to help nursing students acquire and retain knowledge about basic and advanced life support techniques. Nurse Educ Pract. 2021 Jan;50:102961. doi: 10.1016/j.nepr.2020.102961. Epub 2020 Dec 29. PMID 33421681
- [Result] Gutierrez-Puertas L, Marquez-Hernandez VV, Gutierrez-Puertas V, Rodriguez-Garcia MC, Garcia-Viola A, Aguilera-Manrique G. Are You Prepared to Save a Life? Nursing Students' Experience in Advanced Life Support Practice. Int J Environ Res Public Health. 2021 Jan 31;18(3):1273. doi: 10.3390/ijerph18031273. PMID 33572616
- [Result] Haider AS, Al-Salman S. Dataset of Jordanian university students' psychological health impacted by using e-learning tools during COVID-19. Data Brief. 2020 Jul 31;32:106104. doi: 10.1016/j.dib.2020.106104. eCollection 2020 Oct. PMID 32789158
- [Result] Handeland JA, Prinz A, Ekra EMR, Fossum M. The role of manikins in nursing students' learning: A systematic review and thematic metasynthesis. Nurse Educ Today. 2021 Mar;98:104661. doi: 10.1016/j.nedt.2020.104661. Epub 2020 Nov 12. PMID 33298327
- [Result] Higgins BV, Medvedev MM, Spindler H, Ghosh R, Longkumer O, Cohen SR, Das A, Gore A, Mahapatra T, Walker DM. Cohort study of neonatal resuscitation skill retention in frontline healthcare facilities in Bihar, India, after PRONTO simulation training. BMJ Paediatr Open. 2020 Apr 20;4(1):e000628. doi: 10.1136/bmjpo-2019-000628. eCollection 2020. PMID 32399505
- [Result] Holm A, Jerkeman M, Sultanian P, Lundgren P, Ravn-Fischer A, Israelsson J, Giesecke J, Herlitz J, Rawshani A. Cohort study of the characteristics and outcomes in patients with COVID-19 and in-hospital cardiac arrest. BMJ Open. 2021 Nov 30;11(11):e054943. doi: 10.1136/bmjopen-2021-054943. PMID 34848525
- [Result] Irfan B, Zahid I, Khan MS, Khan OAA, Zaidi S, Awan S, Bilal S, Irfan O. Current state of knowledge of basic life support in health professionals of the largest city in Pakistan: a cross-sectional study. BMC Health Serv Res. 2019 Nov 21;19(1):865. doi: 10.1186/s12913-019-4676-y. PMID 31752855
- [Result] Iserbyt P, Theys L, Ward P, Charlier N. The effect of a specialized content knowledge workshop on teaching and learning Basic Life Support in elementary school: A cluster randomized controlled trial. Resuscitation. 2017 Mar;112:17-21. doi: 10.1016/j.resuscitation.2016.11.023. Epub 2016 Dec 20. PMID 28011290
- [Result] Jang K, Kim SH, Oh JY, Mun JY. Effectiveness of self-re-learning using video recordings of advanced life support on nursing students' knowledge, self-efficacy, and skills performance. BMC Nurs. 2021 Mar 31;20(1):52. doi: 10.1186/s12912-021-00573-8. PMID 33789625
- [Result] Jarrah S, Judeh M, AbuRuz ME. Evaluation of public awareness, knowledge and attitudes towards basic life support: a cross-sectional study. BMC Emerg Med. 2018 Oct 29;18(1):37. doi: 10.1186/s12873-018-0190-5. PMID 30373529
- [Result] Jung D, Lee SH, Kang SJ, Kim JH. Development and evaluation of a clinical simulation for new graduate nurses: A multi-site pilot study. Nurse Educ Today. 2017 Feb;49:84-89. doi: 10.1016/j.nedt.2016.11.010. Epub 2016 Nov 18. PMID 27889583
- [Result] Kei J, Mebust DP. Effects of cardiopulmonary resuscitation on direct versus video laryngoscopy using a mannequin model. Am J Emerg Med. 2021 Dec;50:587-591. doi: 10.1016/j.ajem.2021.09.031. Epub 2021 Sep 20. PMID 34563941
- [Result] Kim CH, Kim TH, Shin SD, Song KJ, Ro YS, Ahn KO, Hong KJ, Lee YJ, Lee EJ, Ha SY. The effect of automatic external defibrillator with a real-time feedback on quality of bystander cardiopulmonary resuscitation: A before-and-after simulation study. Health Soc Care Community. 2019 Sep;27(5):e744-e751. doi: 10.1111/hsc.12800. Epub 2019 Jun 21. PMID 31225932
- [Result] Kim YH, Jang KS. [Effect of a simulation-based education on cardio-pulmonary emergency care knowledge, clinical performance ability and problem solving process in new nurses]. J Korean Acad Nurs. 2011 Apr;41(2):245-55. doi: 10.4040/jkan.2011.41.2.245. Korean. PMID 21551996
- [Result] Kose S, Akin S, Mendi O, Goktas S. The effectiveness of basic life support training on nursing students' knowledge and basic life support practices: a non-randomized quasi-experimental study. Afr Health Sci. 2019 Jun;19(2):2252-2262. doi: 10.4314/ahs.v19i2.51. PMID 31656511
- [Result] La Cerra C, Dante A, Caponnetto V, Franconi I, Gaxhja E, Petrucci C, Alfes CM, Lancia L. Effects of high-fidelity simulation based on life-threatening clinical condition scenarios on learning outcomes of undergraduate and postgraduate nursing students: a systematic review and meta-analysis. BMJ Open. 2019 Feb 22;9(2):e025306. doi: 10.1136/bmjopen-2018-025306. PMID 30798316
- [Result] Laco RB, Stuart WP. Simulation-Based Training Program to Improve Cardiopulmonary Resuscitation and Teamwork Skills for the Urgent Care Clinic Staff. Mil Med. 2022 May 3;187(5-6):e764-e769. doi: 10.1093/milmed/usab198. PMID 34050365
- [Result] Lauridsen KG, Morgan RW, Dewan M, Gawronski O, Sen AI; PediRES-Q Investigators. In-hospital cardiac arrest characteristics, CPR quality, and outcomes in children with COVID-19. Resuscitation. 2021 Dec;169:39-40. doi: 10.1016/j.resuscitation.2021.10.013. Epub 2021 Oct 18. No abstract available. PMID 34673154
- [Result] Lee DK. Alternatives to P value: confidence interval and effect size. Korean J Anesthesiol. 2016 Dec;69(6):555-562. doi: 10.4097/kjae.2016.69.6.555. Epub 2016 Oct 25. PMID 27924194
- [Result] Liaw SY, Wong LF, Chan SW, Ho JT, Mordiffi SZ, Ang SB, Goh PS, Ang EN. Designing and evaluating an interactive multimedia Web-based simulation for developing nurses' competencies in acute nursing care: randomized controlled trial. J Med Internet Res. 2015 Jan 12;17(1):e5. doi: 10.2196/jmir.3853. PMID 25583029
- [Result] Magill N, Knight R, McCrone P, Ismail K, Landau S. A scoping review of the problems and solutions associated with contamination in trials of complex interventions in mental health. BMC Med Res Methodol. 2019 Jan 7;19(1):4. doi: 10.1186/s12874-018-0646-z. PMID 30616508
- [Result] Manolis AS, Manolis AA, Manolis TA, Apostolopoulos EJ, Papatheou D, Melita H. COVID-19 infection and cardiac arrhythmias. Trends Cardiovasc Med. 2020 Nov;30(8):451-460. doi: 10.1016/j.tcm.2020.08.002. Epub 2020 Aug 16. PMID 32814095
- [Result] Marijon E, Karam N, Jost D, Perrot D, Frattini B, Derkenne C, Sharifzadehgan A, Waldmann V, Beganton F, Narayanan K, Lafont A, Bougouin W, Jouven X. Out-of-hospital cardiac arrest during the COVID-19 pandemic in Paris, France: a population-based, observational study. Lancet Public Health. 2020 Aug;5(8):e437-e443. doi: 10.1016/S2468-2667(20)30117-1. Epub 2020 May 27. PMID 32473113
- [Result] Maxwell WD, Mohorn PL, Haney JS, Phillips CM, Lu ZK, Clark K, Corboy A, Ragucci KR. Impact of an Advanced Cardiac Life Support Simulation Laboratory Experience on Pharmacy Student Confidence and Knowledge. Am J Pharm Educ. 2016 Oct 25;80(8):140. doi: 10.5688/ajpe808140. PMID 27899836
- [Result] McKelvin R, McKelvin G. Immersive simulation training: Comparing the impact on midwifery and paramedic students' confidence to perform basic life support skills. Midwifery. 2020 Aug;87:102717. doi: 10.1016/j.midw.2020.102717. Epub 2020 Apr 12. PMID 32353663
- [Result] Mendez-Martinez C, Martinez-Isasi S, Garcia-Suarez M, Pena-Rodriguez MA, Gomez-Salgado J, Fernandez-Garcia D. Acquisition of Knowledge and Practical Skills after a Brief Course of BLS-AED in First-Year Students in Nursing and Physiotherapy at a Spanish University. Int J Environ Res Public Health. 2019 Mar 3;16(5):766. doi: 10.3390/ijerph16050766. PMID 30832439
- [Result] Mentzelopoulos SD, Couper K, Voorde PV, Druwe P, Blom M, Perkins GD, Lulic I, Djakow J, Raffay V, Lilja G, Bossaert L. European Resuscitation Council Guidelines 2021: Ethics of resuscitation and end of life decisions. Resuscitation. 2021 Apr;161:408-432. doi: 10.1016/j.resuscitation.2021.02.017. Epub 2021 Mar 24. PMID 33773832
- [Result] Muflih S, Abuhammad S, Al-Azzam S, Alzoubi KH, Muflih M, Karasneh R. Online learning for undergraduate health professional education during COVID-19: Jordanian medical students' attitudes and perceptions. Heliyon. 2021 Sep;7(9):e08031. doi: 10.1016/j.heliyon.2021.e08031. Epub 2021 Sep 20. PMID 34568607
- [Result] Nabolsi M, Abu-Moghli F, Khalaf I, Zumot A, Suliman W. Nursing Faculty Experience With Online Distance Education During COVID-19 Crisis: A Qualitative Study. J Prof Nurs. 2021 Sep-Oct;37(5):828-835. doi: 10.1016/j.profnurs.2021.06.002. Epub 2021 Jun 9. PMID 34742511
- [Result] Nassar AK, Al-Manaseer F, Knowlton LM, Tuma F. Virtual reality (VR) as a simulation modality for technical skills acquisition. Ann Med Surg (Lond). 2021 Oct 27;71:102945. doi: 10.1016/j.amsu.2021.102945. eCollection 2021 Nov. PMID 34840738
- [Result] Nishiyama C, Iwami T, Murakami Y, Kitamura T, Okamoto Y, Marukawa S, Sakamoto T, Kawamura T. Effectiveness of simplified 15-min refresher BLS training program: a randomized controlled trial. Resuscitation. 2015 May;90:56-60. doi: 10.1016/j.resuscitation.2015.02.015. Epub 2015 Feb 24. PMID 25724354
- [Result] Oermann MH, Krusmark MA, Kardong-Edgren S, Jastrzembski TS, Gluck KA. Training interval in cardiopulmonary resuscitation. PLoS One. 2020 Jan 16;15(1):e0226786. doi: 10.1371/journal.pone.0226786. eCollection 2020. PMID 31945074
- [Result] Oteir AO, Almhdawi KA, Kanaan SF, Alwidyan MT, Williams B. Cardiopulmonary resuscitation level of knowledge among allied health university students in Jordan: a cross-sectional study. BMJ Open. 2019 Nov 19;9(11):e031725. doi: 10.1136/bmjopen-2019-031725. PMID 31748305
- [Result] Paddock A. Using Simulation to Improve Adherence to Get With the Guidelines Time to First Shock. Crit Care Nurse. 2021 Dec 1;41(6):62-68. doi: 10.4037/ccn2021596. PMID 34851386
- [Result] Paliatsiou S, Xanthos T, Wyllie J, Volaki P, Sokou R, Bikouli D, Iliodromiti Z, Boutsikou T, Iacovidou N. Theoretical knowledge and skill retention 3 and 6 months after a European Newborn Life Support provider course. Am J Emerg Med. 2021 Nov;49:83-88. doi: 10.1016/j.ajem.2021.05.048. Epub 2021 May 20. PMID 34089968
- [Result] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Result] Parikh P, Samraj R, Ogbeifun H, Sumbel L, Brimager K, Alhendy M, McElroy J, Whitt D, Henderson C, Bhalala U. Simulation-Based Training in High-Quality Cardiopulmonary Resuscitation Among Neonatal Intensive Care Unit Providers. Front Pediatr. 2022 Mar 9;10:808992. doi: 10.3389/fped.2022.808992. eCollection 2022. PMID 35356440
- [Result] Parsons JR, Crichlow A, Ponnuru S, Shewokis PA, Goswami V, Griswold S. Filling the Gap: Simulation-based Crisis Resource Management Training for Emergency Medicine Residents. West J Emerg Med. 2018 Jan;19(1):205-210. doi: 10.5811/westjem.2017.10.35284. Epub 2017 Dec 14. PMID 29383082
- [Result] Partiprajak S, Thongpo P. Retention of basic life support knowledge, self-efficacy and chest compression performance in Thai undergraduate nursing students. Nurse Educ Pract. 2016 Jan;16(1):235-41. doi: 10.1016/j.nepr.2015.08.012. Epub 2015 Sep 3. PMID 26553101
- [Result] Pehlivan M, Mercan NC, Cinar I, Elmali F, Soyoz M. The evaluation of laypersons awareness of basic life support at the university in Izmir. Turk J Emerg Med. 2019 Jan 18;19(1):26-29. doi: 10.1016/j.tjem.2018.11.002. eCollection 2019 Jan. PMID 30793062
- [Result] Perkins GD, Couper K. COVID-19: long-term effects on the community response to cardiac arrest? Lancet Public Health. 2020 Aug;5(8):e415-e416. doi: 10.1016/S2468-2667(20)30134-1. Epub 2020 May 27. No abstract available. PMID 32473112
- [Result] Piryani RM, Piryani S, Shrestha U, Acharya A, Kanskar S, Shahi M, Kayastha J, Chaulagain A, Agarwal JP, Bajracharya SR. Simulation-based education workshop: perceptions of participants. Adv Med Educ Pract. 2019 Jul 23;10:547-554. doi: 10.2147/AMEP.S204816. eCollection 2019. PMID 31413653
- [Result] Rajaguru V, Park J. Contemporary Integrative Review in Simulation-Based Learning in Nursing. Int J Environ Res Public Health. 2021 Jan 15;18(2):726. doi: 10.3390/ijerph18020726. PMID 33467730
- [Result] Roedl K, Soffker G, Fischer D, Muller J, Westermann D, Issleib M, Kluge S, Jarczak D. Effects of COVID-19 on in-hospital cardiac arrest: incidence, causes, and outcome - a retrospective cohort study. Scand J Trauma Resusc Emerg Med. 2021 Feb 8;29(1):30. doi: 10.1186/s13049-021-00846-w. PMID 33557923
- [Result] Rushton MA, Drumm IA, Campion SP, O'Hare JJ. The Use of Immersive and Virtual Reality Technologies to Enable Nursing Students to Experience Scenario-Based, Basic Life Support Training-Exploring the Impact on Confidence and Skills. Comput Inform Nurs. 2020 Jun;38(6):281-293. doi: 10.1097/CIN.0000000000000608. PMID 32149741
- [Result] Ryan A, Rizwan R, Williams B, Benscoter A, Cooper DS, Iliopoulos I. Simulation Training Improves Resuscitation Team Leadership Skills of Nurse Practitioners. J Pediatr Health Care. 2019 May-Jun;33(3):280-287. doi: 10.1016/j.pedhc.2018.09.006. Epub 2018 Nov 27. PMID 30497891
- [Result] Ryzner DM, Kujath AS. Low-Fidelity Code Blue Simulation on the Orthopaedic Unit. Orthop Nurs. 2018 Jul/Aug;37(4):230-234. doi: 10.1097/NOR.0000000000000475. PMID 30028424
- [Result] Saramma PP, Raj LS, Dash PK, Sarma PS. Assessment of long-term impact of formal certified cardiopulmonary resuscitation training program among nurses. Indian J Crit Care Med. 2016 Apr;20(4):226-32. doi: 10.4103/0972-5229.180043. PMID 27303137
- [Result] Sarvan S, Efe E. The effect of neonatal resuscitation training based on a serious game simulation method on nursing students' knowledge, skills, satisfaction and self-confidence levels: A randomized controlled trial. Nurse Educ Today. 2022 Apr;111:105298. doi: 10.1016/j.nedt.2022.105298. Epub 2022 Feb 8. PMID 35158135
- [Result] Sawyer T, Eppich W, Brett-Fleegler M, Grant V, Cheng A. More Than One Way to Debrief: A Critical Review of Healthcare Simulation Debriefing Methods. Simul Healthc. 2016 Jun;11(3):209-17. doi: 10.1097/SIH.0000000000000148. PMID 27254527
- [Result] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Result] Perkins GD, Graesner JT, Semeraro F, Olasveengen T, Soar J, Lott C, Van de Voorde P, Madar J, Zideman D, Mentzelopoulos S, Bossaert L, Greif R, Monsieurs K, Svavarsdottir H, Nolan JP; European Resuscitation Council Guideline Collaborators. European Resuscitation Council Guidelines 2021: Executive summary. Resuscitation. 2021 Apr;161:1-60. doi: 10.1016/j.resuscitation.2021.02.003. Epub 2021 Mar 24. PMID 33773824
- [Result] Sherwood RJ, Francis G. The effect of mannequin fidelity on the achievement of learning outcomes for nursing, midwifery and allied healthcare practitioners: Systematic review and meta-analysis. Nurse Educ Today. 2018 Oct;69:81-94. doi: 10.1016/j.nedt.2018.06.025. Epub 2018 Jun 30. PMID 30015220
- [Result] Shorey S, Pereira TL, Teo WZ, Ang E, Lau TC, Samarasekera DD. Navigating nursing curriculum change during COVID-19 pandemic: A systematic review and meta-synthesis. Nurse Educ Pract. 2022 Nov;65:103483. doi: 10.1016/j.nepr.2022.103483. Epub 2022 Oct 27. PMID 36327596
- [Result] Shrestha R, Badyal D, Shrestha AP, Shrestha A. In-situ Simulation-Based Module to Train Interns in Resuscitation Skills During Cardiac Arrest. Adv Med Educ Pract. 2020 Apr 8;11:271-285. doi: 10.2147/AMEP.S246920. eCollection 2020. PMID 32308520
- [Result] Sindiani AM, Obeidat N, Alshdaifat E, Elsalem L, Alwani MM, Rawashdeh H, Fares AS, Alalawne T, Tawalbeh LI. Distance education during the COVID-19 outbreak: A cross-sectional study among medical students in North of Jordan. Ann Med Surg (Lond). 2020 Nov;59:186-194. doi: 10.1016/j.amsu.2020.09.036. Epub 2020 Oct 2. PMID 33042535
- [Result] Sorensen JL, Ostergaard D, LeBlanc V, Ottesen B, Konge L, Dieckmann P, Van der Vleuten C. Design of simulation-based medical education and advantages and disadvantages of in situ simulation versus off-site simulation. BMC Med Educ. 2017 Jan 21;17(1):20. doi: 10.1186/s12909-016-0838-3. PMID 28109296
- [Result] Staerk M, Vammen L, Andersen CF, Krogh K, Lofgren B. Basic life support skills can be improved among certified basic life support instructors. Resusc Plus. 2021 Apr 14;6:100120. doi: 10.1016/j.resplu.2021.100120. eCollection 2021 Jun. PMID 34223379
- [Result] Suliman WA, Abu-Moghli FA, Khalaf I, Zumot AF, Nabolsi M. Experiences of nursing students under the unprecedented abrupt online learning format forced by the national curfew due to COVID-19: A qualitative research study. Nurse Educ Today. 2021 May;100:104829. doi: 10.1016/j.nedt.2021.104829. Epub 2021 Feb 27. PMID 33740705
- [Result] Tawalbeh LI, Tubaishat A. Effect of simulation on knowledge of advanced cardiac life support, knowledge retention, and confidence of nursing students in Jordan. J Nurs Educ. 2014 Jan 1;53(1):38-44. doi: 10.3928/01484834-20131218-01. Epub 2013 Dec 18. PMID 24328248
- [Result] Teoh SE, Masuda Y, Tan DJH, Liu N, Morrison LJ, Ong MEH, Blewer AL, Ho AFW. Impact of the COVID-19 pandemic on the epidemiology of out-of-hospital cardiac arrest: a systematic review and meta-analysis. Ann Intensive Care. 2021 Dec 7;11(1):169. doi: 10.1186/s13613-021-00957-8. PMID 34874498
- [Result] Thompson Bastin ML, Cook AM, Flannery AH. Use of simulation training to prepare pharmacy residents for medical emergencies. Am J Health Syst Pharm. 2017 Mar 15;74(6):424-429. doi: 10.2146/ajhp160129. PMID 28274986
- [Result] Torsy T, Deswarte W, Karlberg Traav M, Beeckman D. Effect of a dynamic mattress on chest compression quality during cardiopulmonary resuscitation. Nurs Crit Care. 2022 Mar;27(2):275-281. doi: 10.1111/nicc.12631. Epub 2021 Apr 21. PMID 33884701
- [Result] Toubasi S, Alosta MR, Darawad MW, Demeh W. Impact of simulation training on Jordanian nurses' performance of basic life support skills: A pilot study. Nurse Educ Today. 2015 Sep;35(9):999-1003. doi: 10.1016/j.nedt.2015.03.017. Epub 2015 Apr 16. PMID 25935665
- [Result] Umuhoza C, Chen L, Unyuzumutima J, McCall N. Impact of structured basic life-support course on nurses' cardiopulmonary resuscitation knowledge and skills: Experience of a paediatric department in low-resource country. Afr J Emerg Med. 2021 Sep;11(3):366-371. doi: 10.1016/j.afjem.2021.03.014. Epub 2021 Jul 22. PMID 34367898
- [Result] Uzen Cura S, Kocatepe V, Yildirim D, Kucukakgun H, Atay S, Unver V. Examining Knowledge, Skill, Stress, Satisfaction, and Self-Confidence Levels of Nursing Students in Three Different Simulation Modalities. Asian Nurs Res (Korean Soc Nurs Sci). 2020 Aug;14(3):158-164. doi: 10.1016/j.anr.2020.07.001. Epub 2020 Jul 9. PMID 32653666
- [Result] Van de Voorde P, Turner NM, Djakow J, de Lucas N, Martinez-Mejias A, Biarent D, Bingham R, Brissaud O, Hoffmann F, Johannesdottir GB, Lauritsen T, Maconochie I. European Resuscitation Council Guidelines 2021: Paediatric Life Support. Resuscitation. 2021 Apr;161:327-387. doi: 10.1016/j.resuscitation.2021.02.015. Epub 2021 Mar 24. PMID 33773830
- [Result] Waldner MH, Olson JK. Taking the patient to the classroom: applying theoretical frameworks to simulation in nursing education. Int J Nurs Educ Scholarsh. 2007;4:Article18. doi: 10.2202/1548-923X.1317. Epub 2007 Sep 17. PMID 17910532
- [Result] Williams KL, Rideout J, Pritchett-Kelly S, McDonald M, Mullins-Richards P, Dubrowski A. Mock Code: A Code Blue Scenario Requested by and Developed for Registered Nurses. Cureus. 2016 Dec 23;8(12):e938. doi: 10.7759/cureus.938. PMID 28123919
- [Result] Wilson C, Furness E, Proctor L, Sweetman G, Hird K. A randomised trial of the effectiveness of instructor versus automated manikin feedback for training junior doctors in life support skills. Perspect Med Educ. 2021 Mar;10(2):95-100. doi: 10.1007/s40037-020-00631-y. Epub 2020 Nov 26. PMID 33242153
- [Result] Wyckoff MH, Singletary EM, Soar J, Olasveengen TM, Greif R, Liley HG, Zideman D, Bhanji F, Andersen LW, Avis SR, Aziz K, Bendall JC, Berry DC, Borra V, Bottiger BW, Bradley R, Bray JE, Breckwoldt J, Carlson JN, Cassan P, Castren M, Chang WT, Charlton NP, Cheng A, Chung SP, Considine J, Costa-Nobre DT, Couper K, Dainty KN, Davis PG, de Almeida MF, de Caen AR, de Paiva EF, Deakin CD, Djarv T, Douma MJ, Drennan IR, Duff JP, Eastwood KJ, El-Naggar W, Epstein JL, Escalante R, Fabres JG, Fawke J, Finn JC, Foglia EE, Folke F, Freeman K, Gilfoyle E, Goolsby CA, Grove A, Guinsburg R, Hatanaka T, Hazinski MF, Heriot GS, Hirsch KG, Holmberg MJ, Hosono S, Hsieh MJ, Hung KKC, Hsu CH, Ikeyama T, Isayama T, Kapadia VS, Kawakami MD, Kim HS, Kloeck DA, Kudenchuk PJ, Lagina AT, Lauridsen KG, Lavonas EJ, Lockey AS, Malta Hansen C, Markenson D, Matsuyama T, McKinlay CJD, Mehrabian A, Merchant RM, Meyran D, Morley PT, Morrison LJ, Nation KJ, Nemeth M, Neumar RW, Nicholson T, Niermeyer S, Nikolaou N, Nishiyama C, O'Neil BJ, Orkin AM, Osemeke O, Parr MJ, Patocka C, Pellegrino JL, Perkins GD, Perlman JM, Rabi Y, Reynolds JC, Ristagno G, Roehr CC, Sakamoto T, Sandroni C, Sawyer T, Schmolzer GM, Schnaubelt S, Semeraro F, Skrifvars MB, Smith CM, Smyth MA, Soll RF, Sugiura T, Taylor-Phillips S, Trevisanuto D, Vaillancourt C, Wang TL, Weiner GM, Welsford M, Wigginton J, Wyllie JP, Yeung J, Nolan JP, Berg KM; COVID-19 Working Group. 2021 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations: Summary From the Basic Life Support; Advanced Life Support; Neonatal Life Support; Education, Implementation, and Teams; First Aid Task Forces; and the COVID-19 Working Group. Resuscitation. 2021 Dec;169:229-311. doi: 10.1016/j.resuscitation.2021.10.040. Epub 2021 Nov 11. PMID 34933747
- [Result] Zideman DA, Singletary EM, Borra V, Cassan P, Cimpoesu CD, De Buck E, Djarv T, Handley AJ, Klaassen B, Meyran D, Oliver E, Poole K. European Resuscitation Council Guidelines 2021: First aid. Resuscitation. 2021 Apr;161:270-290. doi: 10.1016/j.resuscitation.2021.02.013. Epub 2021 Mar 24. PMID 33773828
- [Derived] Abu-Wardeh Y, Ahmad WMAW, Che Hamzah MSS, Najjar YW, Hassan II. Enriching nursing knowledge and practice in Jordanian government hospitals through basic life support simulation training: A randomized controlled trial. Belitung Nurs J. 2024 Jun 28;10(3):261-271. doi: 10.33546/bnj.3328. eCollection 2024. PMID 38947304
- See also: The Effect of Medium Fidelity Simulation on Perceived Competence Level of Novice Nursing Students — http://search.ebscohost.com/login.aspx?direct=true&db=jlh&AN=109860356&lang=es&site=ehost-live
- See also: Effects of in-situ simulation training intervention on Intensive Care Unit and Emergency Department nurses ' competency and confidence to ability to perform cardio- pulmonary resuscitation — https://www.theseus.fi/handle/10024/227686
- See also: Descriptive comparative study of nursing faculty self-efficacy in the simulation setting. Descriptive Comparative Study of Nursing Faculty Self-Efficacy in the Simulation Setting — http://lib.tcu.edu/PURL/EZproxy_link.asp?url=https://search.ebscohost.com/login.aspx?direct=true&AuthType=cookie,ip,uid&db=ccm&AN=123295984&site=ehost-live
- See also: Brown, D. K., & Benson, S. N. K. (2020). Does Time in Team Training Matter ? Evaluation of Team-Level Attitudes With Interprofessional Education. Clinical Simulation in Nursing, 48, 38-45 — https://doi.org/10.1016/j.ecns.2020.08.002
- See also: To assess the effectiveness of simulation teaching of defibrillation on the knowledge and skill of nurses working in the critical care unit of a Tertiary Care Teaching Institute: Prospective, — https://doi.org/10.4103/ijcn.ijcn_31_20
- See also: The Effects of Repeated Basic Life Support Training on Teachers' Knowledge and Skill Levels: A Quasi-experimental Study. Eurasian Journal of Emergency Medicine, 19(1), 46-51 — https://doi.org/10.4274/eajem.galenos.2019.47450
- See also: A Study on How Beneficial Simulation Experience Is For Nursing Staff's Advanced Cardiac Life Support Knowledge at the New Najran General Hospita. Annals of Case Reports, 6(02) — https://doi.org/10.29011/2574-7754.100596
- See also: Purposeful Simulation Role Assignment. Clinical Simulation in Nursing — https://doi.org/10.1016/j.ecns.2020.07.008
- See also: Exploring nurses' knowledge of basic life support guideline of american heart association: A local study. Journal of Emergency Practice and Trauma — https://doi.org/10.34172/jept.2021.02
- See also: Knowledge and Practice of Basic Life Support ( BLS ) Among Registered Nurse at a Private Hospital in Seremban. 13(January), 58-64 — https://doi.org/10.31674/mjn.2022.v13i03.009
- See also: Jawabreh, N., Ayed, A., & Batran, A. (2019). Effect of High Fidelity Simulation on Nursing Students' Knowledge in Palestine. Open Journal of Nursing, 09(04), 364-369 — https://doi.org/10.4236/ojn.2019.94033
- See also: Deliberate Practice in Simulation : Evaluation of Repetitive Code Training on Nursing Students ' BLS Team Skills. Clinical Simulation in Nursing, 48, 8-14 — https://doi.org/10.1016/j.ecns.2020.08.001
- See also: High Fidelity Simulation Experience and Development of Clinical Judgment: Recent Graduate Nurses' Reflections. ProQuest Dissertations and Theses, 127. — https://manchester.idm.oclc.org/login?url=https://search.proquest.com/docview/2070939340?accountid=12253%0Ahttp://man-fe.hosted.exlibrisgroup.com/openurl/44MAN/44MAN_services_page?genre=dissertations+%26+theses&atitle=&author=Lawrence%2C+Martha+Kay&volume
- See also: Quality improvement for self-confidence, critical-thinking, and psychomotor skills in basic life support of nursing health professionals through case-scenario simulation training. Journal of Nursing Education — https://doi.org/10.5430/jnep.v11n8p23
- See also: Guidance for Comprehensive Health Care Simulation Program Evaluation. Clinical Simulation in Nursing, 48, 20-28 — https://doi.org/10.1016/j.ecns.2020.08.003
- See also: Mcdermott, D. S., & Ludlow, J. (2022). A Prebriefing Guide for Online , Virtual , or Distant Simulation Experiences. Clinical Simulation in Nursing, 67, 1-5. — https://doi.org/10.1016/j.ecns.2022.03.004
- See also: Assessing ventilation skills by nursing students in paediatric and adult basic life support: A crossover randomized simulation study using Bag-Val — https://doi.org/10.22514/sv.2020.16.0072
- See also: In Situ Simulation : Challenges and Results (Vol.3: Performance and Tools). Approaches in Patient Safety: New Directions and Alternative Approaches, 1-18 — https://www.ncbi.nlm.nih.gov/books/NBK43682/pdf/Bookshelf_NBK43682.pdf
- See also: A study to assess knowledge andpractice of basic life support among nurses working in tertiary care hospital, New Delhi, India. Nursing & Care Open Access Journal, 7(2), 48-52. — https://doi.org/10.15406/ncoaj.2020.07.00217
- See also: Assessment of the knowledge level and its relevance in terms of CPR in medical personnel of the hospital emergency medical system of the Autonomous Community of the Region of Murcia — https://doi.org/10.6018/eglobal.14.3.197791
- See also: The additional ımpact of simulation based medical training to traditional medical training alone in advanced cardiac life support: A scenario based evaluation — https://doi.org/10.22514/SV142.102018.10
- See also: Atualização de trabalhadores de enfermagem em suporte básico de vida. Revista de Enfermagem UFPE on Line, 13 — https://doi.org/10.5205/1981-8963.2019.241981
- See also: The Effect of High-Fidelity Cardiopulmonary Resuscitation (CPR) Simulation on Athletic Training Student Knowledge, Confidence, Emotions, and Experiences. Athletic Training Education Journal, 10(2), 103-112. — https://doi.org/10.4085/1002103
- See also: Suporte básico de vida: Avaliação da aprendizagem com uso de simulação e dispositivos de feedback imediato. Revista Latino-Americana de Enfermagem — https://doi.org/10.1590/1518-8345.1957.2942
- See also: Knowledge Level of Healthcare Professionals on Basic and Advanced Life Support in Children. Eurasian Journal of Emergency Medicine — https://doi.org/10.4274/eajem.galenos.2020.05579
- See also: Resuscitation and Emergency Cardiovascular Care Aid Task Forces ; and the COVID-19 Working Group International Liaison Committee on Resuscitation. 9. https://doi.org/10.1016/j.resuscitation.2021.10.040 — https://doi.org/10.1016/j.resuscitation.2021.10.040
- See also: Knowledge, attitude and practice of basic life support among junior doctors and students in a tertiary care medical institute. International Journal of Research in Medical Sciences — https://doi.org/10.18203/2320-6012.ijrms20151416
- See also: High Fidelity Simulation Improves Provider Confidence During ACLS Training Even Among Experienced Staff: Are We Missing an Opportunity? Emergency Medicine — https://doi.org/10.17140/emoj-2-120

DOCUMENTS (3):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06001879/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06001879/SAP_001.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06001879/ICF_002.pdf